CLINICAL TRIAL: NCT03925818
Title: Twice-a-day PPI, Tetracycline, Metronidazolequadruple Therapy With Pylera® or Lactobacillus Reuteri for Treatment naïve or for Retreatment of H. Pylori: Two Randomized Pilot Studies
Brief Title: Low Dose Bismuth Versus Lactobacillus Reuteri for H. Pylori Eradication
Acronym: LactoBismu
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lactobacillus reuteri (Gastrus®) was not anymore available in the region
Sponsor: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, Maria Pina Dore, Professor, Università degli Studi di Sassari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2358/CE
Record Dates: First submitted 2019-04-19; First posted 2019-04-24 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Helicobacter Pylori Infection
Keywords: Lactobacillus reuteri; Bismuth; Helicobacter pylori;
MeSH Terms: interventions — Metronidazole; Tetracycline; Pantoprazole; Bismuth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B.I.D. TMPPI + Lactobacillus-10 (Experimental): pantoprazole 20 mg, tetracycline 500 mg, and metronidazole 500 mg twice a day supplemented with 1 capsule (2 x 108 CFU of L. reuteri DSM 17938 plus 2 x 108 CFU of L. reuteri ATCC PTA 6475) a day in the afternoon, given with the midday and evening meals for 10 days
  Interventions: Drug: Bismuth Subcitrate Potassium
- B.I.D. Bismuth (Active Comparator): pantoprazole 20 mg and the same doses of antibiotics administered as tetracycline 250 mg, and metronidazole 250 mg plus 1 cp (140 mg bismuth subcitrate potassium, 125 mg metronidazole, and 125 mg tetracycline hydrochloride administered) x 2 all drugs twice-a-day given with the midday and evening meals for 10 days
  Interventions: Dietary Supplement: Gastrus

INTERVENTIONS:
Drug: Bismuth Subcitrate Potassium — Pylera capsules
  Other Names: Pylera; Metronidazole, Tetracycline, pantoprazole, Bismuth
  Arms: B.I.D. TMPPI + Lactobacillus-10
Dietary Supplement: Gastrus — Gastrus 1 tablet
  Other Names: L. reuteri DSM 17938 and L. reuteri ATCC PTA 6475
  Arms: B.I.D. Bismuth

SUMMARY:
This study investigates the efficacy of a b.i.d. quadruple therapy containing Pylera® or L. reuteri for H. pylori infection.

DETAILED DESCRIPTION:
Bismuth, metronidazole and tetracycline yielded high cure rates for H. pylori infection. Earlier studies suggested that the bismuth quadruple therapy may be effective when given twice-a-day rather than q.i.d. and that b.i.d. therapy was associated with fewer side effects. The addition of the probiotic Lactobacillus reuteri (Gastrus®) to Lactobacillus reuteri (Gastrus®) that has been shown to increase the cure rates by 10-14%. In another study bismuth supplementation with L. reuteri DSM 17938, in a modified low dose quadruple therapy provided good eradication rates (93.3%; 95% CI : 85-99%) in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

- Positive for H. pylori infection

Exclusion Criteria:

* Presence of malignancy
* Pregnancy or lactation
* Clinically significant diseases
* History of drug or alcohol abuse
* Allergy to pantoprazole or to any component of regimens used in the study
* Use of anti-secretory drugs, antibiotics or probiotics 4 weeks preceding the enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2018-12-23 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | 30-40 days after the end of treatment
  a negative 13C-urea breath test and/or a negative stool antigen test

SECONDARY OUTCOMES:
Compliance and side effects evaluation | 30-40 days
  Patient interview at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: MARIA P Dore, MD, PhD, Principal Investigator — Università degli Studi di Sassari
Locations (1):
- Clinica Medica, Dipartimento di Medicina Clinica e Sperimentale, Sassari, SS, Italy